CLINICAL TRIAL: NCT06334315
Title: Influence of Genetics Variants on the Pharmacokinetics and Pharmacodynamics of Combined Oral Contraceptive Pill Users
Brief Title: Oral Contraceptive Pill (OCP) Pharmacogenomics
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000037337; R01HD111436 (NIH)
Record Dates: First submitted 2024-03-13; First posted 2024-03-28 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Contraception; Pharmacogenomic Drug Interaction
MeSH Terms: interventions — Desogestrel; Ethinyl Estradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Combined oral contraceptive pill users (Experimental): Administered a combined oral contraceptive pill containing desogestrel and ethinyl estradiol (Desogen, 0.15mg desogestrel and 0.03mg ethinyl estradiol per active pill) for at least one cycle (21 days) and up to 13 total cycles (one year)
  Interventions: Drug: Desogestrel / Ethinyl Estradiol Pill

INTERVENTIONS:
Drug: Desogestrel / Ethinyl Estradiol Pill — Standard pill packs containing 21 active pills and 7 placebo pills

SUMMARY:
The goal of this clinical trial is to evaluate how differences in specific parts of our DNA can influence how individual bodies break down the hormones contained within oral contraceptive pills, which could affect how well these birth control pills work to prevent pregnancy. The investigators are also interested in exploring how these differences in our DNA can also explain why patients taking the exact same formulation of birth control pill will experience very different side effects. The main questions it aims to answer are:

* Do individuals with the CYP3A7*1C variant have increased metabolism of both desogestrel and ethinyl estradiol when taking a combined oral contraceptive pill?
* Do individuals with the CYP3A7*1C variant experience higher rates of breakthrough ovulation while taking a desogestrel/ethinyl estradiol combined oral contraceptive pill?
* What novel genetic loci are associated with alterations in steroid hormone pharmacokinetics and pharmacodynamics among a larger cohort of combined oral contraceptive pill users?

Participants will take a specific formulation of combined oral contraceptive pill (desogestrel/ethinyl estradiol) and undergo the following procedures:

* Blood draw to measure the amount of progestin and estrogen in their system from the combined oral contraceptive pill
* Questionnaires to assess side effects possibly caused by the combined oral contraceptive pill
* Blood draw to measure endogenous hormone levels and biomarkers that may be affected by the combined oral contraceptive pill
* A transvaginal ultrasound to measure any ovarian follicles (optional procedure)

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Female, aged 18-45 years old
4. In good general health as evidenced by medical history and no need for regular intensive medical interventions (e.g., inpatient admissions, surgical treatments). The Principal Investigator will be responsible for determining good general health for potential participants with complicated medical histories.
5. Ability to take oral medication and be willing to adhere to the oral contraceptive pill (DSG/EE) regimen
6. Body-mass index ≥18.5kg/m2
7. Willing to abstain from medications and supplements known to induce/inhibit CYP3A (e.g., rifampin, carbamazepine, ketoconazole, St. John's wort) during the study
8. Normal blood pressure measurement at study screening
9. Negative urine pregnancy test at study screening

Exclusion Criteria:

1. Currently taking any known CYP3A inducers/inhibitors (e.g., rifampin, carbamazepine, ketoconazole, St. John's wort)43
2. Any medical conditions that affect liver function (e.g., hepatitis, cirrhosis)
3. Contraindications to estrogen-containing contraception (based on category 3 or 4 recommendations in the CDC MEC guidelines42)

   1. Current breast cancer or personal history of breast cancer
   2. Severe decompensated cirrhosis
   3. Personal history of deep venous thrombosis or pulmonary embolism
   4. Recent major surgery with prolonged immobilization
   5. Diabetes with nephropathy, retinopathy, neuropathy, or other vascular disease
   6. Current gallbladder disease
   7. Migraine headaches with aura
   8. History of malabsorptive bariatric surgery
   9. History of cholestasis due to past oral contraceptive pill use
   10. Personal history of hypertension
   11. Personal history of ischemic heart disease
   12. Known thrombogenic mutations
   13. Personal history of focal nodular hyperplasia of the liver, hepatocellular adenoma, or malignant hepatoma
   14. Multiple sclerosis with prolonged immobility
   15. History of peripartum cardiomyopathy
   16. Current tobacco smoker and age ≥35 years
   17. History of complicated solid organ transplantation
   18. Personal history of stroke
   19. Personal history of superficial venous thrombosis
   20. Systemic lupus erythematosus with positive or unknown antiphospholipid antibodies
   21. Complicated valvular heart disease
   22. Current use of fosamprenavir or lamotrigine
4. Use of injectable contraceptive method within 6 months or current use of an ENG implant
5. Childbirth within 6 months

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 700 (Estimated)
Dates: Start 2024-10-29 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Serum etonogestrel concentration | Measured as a trough concentration on Cycle 1, Day 22 (each cycle is 28 days)
  Pharmacokinetic measurement for progestin
Serum ethinyl estradiol concentration | Measured as a trough concentration on Cycle 1, Day 22 (each cycle is 28 days)
  Pharmacokinetic measurement for estrogen

SECONDARY OUTCOMES:
Serum estradiol concentration | Measured on Cycle 1, Day 22 (all participants), repeated measure in Cycles 3, 6, and 13 (optional study procedures) (each cycle is 28 days)
  Pharmacodynamic measurement of endogenous estrogen
Serum progesterone concentration | Measured on Cycle 1, Day 22 (all participants), repeated measure in Cycles 3, 6, and 13 (optional study procedures) (each cycle is 28 days)
  Pharmacodynamic measurement of endogenous progesterone
Modified Hoogland score | Measured on Cycle 1, Day 22 (optional study procedure) (each cycle is 28 days)
  Calculated based on serum estradiol, serum progesterone, and follicle-like structures. found on transvaginal ultrasound. Scores range from 1 to 5, with a higher score indicating a higher likelihood of pending ovulation with a score of 5 indicating suspected ovulation
Positive and Negative Affect Scheduled | Baseline measured at enrollment, repeat measurement at Cycle 1, Day 22 (all participants), repeated measurements again in Cycles 3, 6, and 13 (optional study procedures) (each cycle is 28 days)
  Questionnaire designed to assess current affect. Scores range from 10-50 for positive affect items and 10-50 for negative affect items, with higher scores representing more positive affect or negative affect, respectively.
Sex hormone binding globulin levels | Baseline measured at enrollment, repeat measurement at Cycle 1, Day 22 (all participants), repeat measurements in cycles 3, 6, and 13 (optional study procedures) (each cycle is 28 days)
  Marker of estrogenicity
Serum albumin concentration | Baseline measured at enrollment, repeat measurement at Cycle 1, Day 22 (all participants), repeat measurements in cycles 3, 6, and 13 (optional study procedures) (each cycle is 28 days)
  Protein binding compound

CONTACTS AND LOCATIONS:
Overall Officials: Aaron M Lazorwitz, MD, PhD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Yale University, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: Yes
IPD will be made available to other researchers at the conclusion of this study and after publication of its findings. Data will be uploaded to dbGaP with individual-level data for genotypes and phenotypes collected in this study.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: De-identified data will be uploaded to dbGaP within one year of completion of the study and will be available indefinitely
Access Criteria: Per dbGaP requirements
URL: https://www.ncbi.nlm.nih.gov/gap/